CLINICAL TRIAL: NCT06604429
Title: Quality of Life Variations Among Adolescent Females Following Virtual Reality Games Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mina Atef Georgui Elias (Other)
Responsible Party: Sponsor-Investigator, Mina Atef Georgui Elias, Lecturer of Physical Therapy, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014233-7; IRB00014233-7 (Other: Faculty of Physical Therapy, Badr University in Cairo)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Obesity-related Medical Conditions; Menstrual Pain; Adolescent Obesity; Body Fat Composition; Obesity; Depression, Anxiety
Keywords: Obesity; Adolescent girls; Body Fat Composition; Menstrual Pain; Virtual reality Games; Aerobic exercise; Diet; Adolescent Obesity; Quality of Life; Depression; Anxiety; Stress; DASS-21
MeSH Terms: conditions — Obesity; Dysmenorrhea; Pediatric Obesity; Depression; Anxiety Disorders | interventions — Exercise; Nutrition Assessment; Exergaming

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exercise (Experimental): The group included 50 girls who received diet advice, aerobic and virtual reality exercises 3 times per week for 8 weeks. they received diet advice and aerobic exercises in form of cycle ergometer training (Each girl started session with a 5 min of warm-up. The exercise phase is performed at 65-75% of age-predicted peak heart rate using an orbitrack device for 20 minutes). Then This was followed by the main part, which consisted of 25 min of exercise when girl immersed in the game and did physical activities for the upper and lower extremities according to the game's requirements, and finally a 5 min cool-down part to lower the heart rate and end the session with static flexibility routines, the total session that would be applied about 50 min (including 30 mins of Virtual reality exercises)
  Interventions: Other: Aerobic exercise; Other: Diet Advice; Other: Virtual reality exercise
- Control group (aerobic exercise) (Active Comparator): This group serves as the control group, it included 50 girls who received diet advice and aerobic exercises in form of cycle ergometer training for 3 times per week for 8 weeks. Each girl started session with a 5 min of warm-up. The exercise phase is performed at 65-75% of age-predicted peak heart rate using an orbitrack device for 20 minutes. Finally, a 5 min cool-down period is permitted, the total session that would be applied about 30 min.
  Interventions: Other: Aerobic exercise; Other: Diet Advice

INTERVENTIONS:
Other: Aerobic exercise — aerobic exercises in form of cycle ergometer training (Each girl started session with a 5 min of warm-up. The exercise phase is performed at 65-75% of age-predicted peak heart rate using an orbitrack device for 20 minutes). Finally, a 5 min cool-down period is permitted, the total session that would be applied about 30 min.
Other: Diet Advice — Adolescent girls participated in the study receive diet advices based on a balanced low calorie diet (1500 Kcal)
Other: Virtual reality exercise — Virtual reality game exercise involves 25 min of exercise where adolescent girl immersed in the game and did physical activities for the upper and lower extremities according to the game's requirements, and finally a 5 min cool-down part to lower the heart rate and end the session with static flexibility routines, the total session that would be applied about 30 min of Virtual reality exercises.
  Arms: Virtual Reality Exercise

SUMMARY:
to compare the effects of virtual reality games, aerobic exercise, and dietary modifications on Quality of Life among adolescent females.

DETAILED DESCRIPTION:
The study will assess whether virtual reality games, aerobic exercise, and dietary modifications lead to significant differences in Quality of Life scores, and perceived exertion as measured by the Borg scale. Additionally, the study will evaluate whether these interventions produce varying impacts on psychological factors such as depression, anxiety, and stress, and on physical measurements like waist circumference (WC) and body fat composition.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescent girls
* Class I Obesity (Body Mass Index from 30 to 34.99 kg/m2)
* Have regular menstruation
* Clinically and medically stable
* no impairment of sensation or other neurological or psychological problems

Exclusion Criteria:

* Visual and/or auditory defects
* Normal weight girls (Body Mass Index from 18 to 24.99 kg/m2) or below average weight (BMI less than 18 kg/m2) or Class II & III Obesity (BMI above 35 kg/m2)
* Girls with significant tightness and/or fixed deformity of lower limbs
* Participants with neurological disorders that affect balance or mentality (e.g. epilepsy).
* Girls with advanced radiographic changes include: Bone destruction, Bony ankylosis, Knee joint subluxation, and Epiphysial fracture)
* Congenital or acquired lower limb deformities in the lower limbs.
* Cardiopulmonary dysfunction.
* Girls under insulin therapy, uncontrolled bronchial asthma, anemia, and Pathological causes of obesity (endocrinal, genetic syndromes...etc.).

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — The study enrolls only biological females and will accept only cisgender girls.
Enrollment: 100 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Body mass index | From enrollment to the end of treatment at 8 weeks
  It is the weight (in kilograms) divided by the height (in meter squares)
Fat Mass | From enrollment to the end of treatment at 8 weeks
  Body fat mass percentage measured by body composition analysis device
Body Water Content | From enrollment to the end of treatment at 8 weeks
  Total body water content percentage measured by body composition analysis device.
Muscle mass | From enrollment to the end of treatment at 8 weeks
  Body muscle mass percentage measured by body composition analysis device.
Waist Circumference | From enrollment to the end of treatment at 8 weeks
  Waist circumference measured in centimeters, where the patient would be in standing position while investigator applied the tape round the abdomen at its narrowest point between the lower rib margin and top of iliac crest at the end of quiet expiration.
Waist hip ratio | From enrollment to the end of treatment at 8 weeks
  It is the ratio between the waist circumference and the hip circumference. Where the waist circumference should be measured at the midpoint between the lower margin of the last palpable ribs and the top of the iliac crest, using a tape measurement. While, the hip circumference should be measured around the widest portion of the buttocks, with the tape parallel to the floor.
Borg Scale (rate of perceived exertion) | From enrollment to the end of treatment at 8 weeks
  This is the modified Borg scale (rating from 0 to 10) where 0 means "no exertion at all" and 20 means "maximal exertion." When a measurement is taken, a number is chosen from the scale by the participant that best describes their perceived level of exertion during physical activity (Six-Minute walk test)

SECONDARY OUTCOMES:
Menstrual pain by Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 8 weeks
  The VAS is a 10-point scale comprising a number from 0 through 10; 0 indicates no pain, and 10 indicates the worst imaginable pain. Adolescent girls participating in the study were instructed to choose a single number from the scale that best indicates their level of menstrual pain
Pediatric Quality of Life Inventory (PedsQL) | From enrollment to the end of treatment at 8 weeks
  It is a 23-item generic health status instrument that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in adolescents.
  The PedsQL 4.0 has been proposed as a valid and reliable generic pediatric HRQOL measurement that can be used for self-reports in age groups ranging from 2 to 18 years and can also be used in clinical practice, clinical trials, and research, as well as school health settings, and community populations.
  It is a questionnaire for the child about child's physical, emotional, social, and school functioning in the past one month. On the PedsQL Generic Core Scales, for ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).
Depression Score | From enrollment to the end of treatment at 8 weeks
  Through the DAAS-21 scale (Depression, Anxiety and Stress scoring and degree)
  It consists of 21 questions, seven questions for depression, seven for anxiety and seven for stress assessment. The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress.
Anxiety Score | From enrollment to the end of treatment at 8 weeks
  Through the DAAS-21 scale (Depression, Anxiety and Stress scoring and degree)
  It consists of 21 questions, seven questions for depression, seven for anxiety and seven for stress assessment. The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress.
Stress Score | From enrollment to the end of treatment at 8 weeks
  Through the DAAS-21 scale (Depression, Anxiety and Stress scoring and degree)
  It consists of 21 questions, seven questions for depression, seven for anxiety and seven for stress assessment. The DASS is a quantitative measure of distress along the 3 axes of depression, anxiety and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Saeed, PhD, Study Chair — Lecturer Dept. of PT for Women's Health Faculty of Physical Therapy Badr University in Cairo, Egypt; Radwa S Abdulrahman, PhD, Principal Investigator — Ass. Prof. Dept. of PT for Pediatric, Faculty of Physical Therapy, Badr University in Cairo, Egypt.; Hayam M Mahmoud, PhD, Study Chair — Professor Dept. of PT for Neurology & Neurosurgery, Faculty of Physical Therapy, Cairo Univ. Egypt.; Wael OA Abd El-Khalek, PhD, Study Chair — Lecturer, Dept. of Basic Sciences, Faculty of Physical Therapy, Badr University in Cairo, Egypt.
Locations (3):
- Egypt (3):
  - Badr University in Cairo faculty of physical therapy, Cairo
  - El-Mahaba Specialized Charity Polyclinics, Cairo
  - Life clinic (Private Clinic) - Minya Al Qamh - Sharqia Governorate, Zagazig